CLINICAL TRIAL: NCT04277767
Title: The Combination of Ophthalmologic Tests and EEG Imaging as a New Biomarker for Alzheimer's Disease
Brief Title: The Role of Ophthalmologic Tests and EEG Imaging in Alzheimer's Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jin Yuan, assistant dean, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: AD2020
Record Dates: First submitted 2020-01-13; First posted 2020-02-20 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Mild Cognitive Impairment
Keywords: AD EEG OCT biomarker
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild cognitive impairment (MCI): observational
  Interventions: Diagnostic Test: observational
- Patients with mild to moderate AD: observational
  Interventions: Diagnostic Test: observational
- Normal controls: observational
  Interventions: Diagnostic Test: observational

INTERVENTIONS:
Diagnostic Test: observational — No intervention

SUMMARY:
Alzheimer's disease (AD) is a prevalent, long-term progressive degenerative disorder with great social impact. It is currently thought that, in addition to neurodegeneration, vascular changes also play a role in the pathophysiology of the disease. Meantime, EEG resting state has also demonstrated significant change in patients with AD in neuroscience research area. Thus, the combination of these sensitive biomarkers would lead to a potential new biomarker for detection of AD, which has higher specificity and sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease

Exclusion Criteria:

* neurologic disorders
* psychiatric disorders

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We would recruit three groups of elders. One is the control group without cognitive impairment, one is the aMCI group which is deemed as the pre-stage of AD, and also the AD group.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
OCT retinal and choroidal thickness | 2 days
  retinal structural anatomy
Retinal Photography vascular caliber | 2 days
  use Retinal Photography to detect vascular caliber
functional connection strength in the brain network | 7 days
  record resting-state EEG, use graph theory to calculate the functional connection strength

CONTACTS AND LOCATIONS:
Overall Officials: Jin Yuan, phD, Principal Investigator — Zhongshan Ophthalmological Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided